CLINICAL TRIAL: NCT04265521
Title: A Prospective Single-arm Investigation to Assess the Efficacy and Safety After Using BioCool Footcare (Footbath) for 3 Weeks of Treatment in Subjects With Mild to Moderate Symptoms/Signs of Tinea Pedis Interdigitalis and Heel Cracks, Calluses and/or Dry Feet.
Brief Title: Study With BioCool Footcare in Subjects With Tinea Pedis Interdigitalis and Heel Cracks, Calluses and/or Dry Feet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biocool AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BioC001
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Foot Fungus; Tinea; Tinea Pedis; Mycoses; Skin Diseases
MeSH Terms: conditions — Tinea; Tinea Pedis; Mycoses; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biocool Footcare (Experimental): Treatment regime:
  During week 1: Once daily for 7 days (7 doses) During week 2 and 3: Once every second day for 14 days (7 doses)
  Interventions: Device: Biocool Footcare

INTERVENTIONS:
Device: Biocool Footcare — BioCool Footcare is a footbath containing granulate of sodium percarbonate that will in this study be used for treatment of foot fungus, heel cracks, calluses and/or dry feet.

SUMMARY:
A prospective, open, post-market study that will enroll male and female subjects diagnosed with foot fungus and at least one of the following conditions: heel cracks, calluses and/or dry feet. The investigation will consist of approximately 48 subjects (considering a 10% drop-out/screening failure rate) fulfilling the eligibility criteria for the study. Each subject will be treated with the study product, BioCool Footcare (footbath), for 3 weeks. The study duration is estimated to 5 months including recruiting, treatment and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

The subjects have to meet all of the following criteria to be eligible to participate in the clinical investigation:

1. Signed informed consent form
2. > 18 years of age
3. Males and females
4. Tinea Pedis (Athlete's foot) confirmed with total symptom score graded between 6-16 (erythema, erosions, macerations, pruritus, fissures, burning/stinging, hyperkeratosis and odour) using a 4-point severity scale (0=absent, 1=mild, 2=moderate and 3=severe). NOTE! maximum total score is 24.

   - Score of 2 (moderate) of higher required in at least 1 of the following; erythema, macerations, pruritus or odur.
5. Score of at least 2 (moderate) required in at least one of the following: heel cracks (rhagades), calluses (hyperkeratosis) and dry feet using a 5-point severity scale (0=absent, 1=mild, 2=moderate, 3=advanced and 4=severe).
6. Patient with confirmed mycological culture

Exclusion Criteria:

Subjects meeting any of the following criteria will not be permitted to participate in the clinical investigation:

1. Severe tinea pedis interdigitalis (Athlete's foot) total score of severity grading >16 (signs and symptoms)
2. Women pregnant or lactation at time of enrolment
3. Diagnosed with Diabetes Type I or II
4. Topical medicinal antifungal therapy within 4 weeks prior to study start
5. Treatment with systemic anti fungal therapy including terbinafine, itraconazole or fluconazole within 6 months prior to study start
6. Treatment with local amd/or systemic corticosteroids or immunosuppressant's within 6 weeks prior to study start
7. Any other open wounds/lesions in the area treated with the Investigational device
8. Participated in another Clinical Investigation/Trial the last 3 months
9. Any other medical condition, judged by the investigator may make follow-up or investigation inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Symptoms of foot fungus | Baseline to end of study (3 weeks)
  Effective treatment rate of the eight clinical signs and symptoms (erythema, erosions, macerations, pruritus, fissures, burning/stinging, hyperkeratosis and odour) using a 4-point severity scale (0=absent, 1=mild, 2=moderate and 3=severe)

SECONDARY OUTCOMES:
Frequency of negative fungual culture in combination with negative KOH test | Baseline to end of study (3 weeks)
  Frequency of subjects with negative fungual culture in combination with negative KOH test
Tolerability assessment to BioCool Footcare (foothbath) | Baseline to end of study (3 weeks)
  Tolerability assessed using a 5-point likert scale (very good, good, moderate, poor, very poor)
Follow-up on heel cracks, calluses and/or dry feet | Baseline to end of study (3 weeks)
  Subject outcome on heel cracks (rhagades), calluses (hyperkeratosis) and/or dry feet using a 5-point scale (0=absent, 1=mild, 2=moderate, 3=advanced, 4=severe)
Dermatology Quality of Life | Baseline to end of study (3 weeks)
  Dermatology Quality of Life Index
Adverse Events | Baseline to end of study (3 weeks)
  Adverse Events (AE, ADE, SAE, SADE, USADE)

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Forskningsenheten Carlanderska sjukhuset, Gothenburg
  - Avdelningen för klinisk prövning, Örebro

IPD SHARING:
Plan to Share IPD: No